# Engagement Trends in Clinical Trials for Metastatic Prostate Cancer - A Journey Into Participation Patterns Among Individuals Affected by the Condition

An Informed Consent Form For Power Clinical Trial's

Observational Study Patients With Metastatic Prostate Cancer

Date: August 18, 2023

Insights into This Informed Consent Document

Should you find yourself tasked with completing this document, it signifies your potential inclusion in an observational clinical trial that specifically addresses individuals having metastatic prostate cancer. This document serves as a comprehensive manual, revealing the study's overarching goals, intricate execution strategy, and diverse implications, both positive and potentially otherwise. Engaging in through contemplation of your prospective participation before making a decision is of paramount importance, and seeking counsel from a trusted advisor can offer invaluable perspectives. In case any aspects of the information contained herein appear ambiguous or if queries arise, be assured that the researcher is readily available to provide clarifications.

# Purpose of the Investigation

Metastatic prostate cancer, also known as advanced or stage IV prostate cancer, is a type of cancer that has originated in the prostate gland and has spread to other parts of the body, usually through the bloodstream or lymphatic system. In metastatic prostate cancer, cancer cells have broken away from the original tumor in the prostate and have established new growths, or metastases, in distant organs or tissues.

Clinical trials aimed at addressing metastatic prostate cancer play a pivotal role in evaluating the safety and efficacy of novel treatments for this condition. These trials are essential in ascertaining whether these emerging treatments surpass current options and provide substantial evidence to support their broader adoption.

This particular study places a meticulous focus on exploring the experiences of individuals diagnosed with metastatic prostate cancer as they actively participate in a unique clinical trial involving medical interventions. The primary emphasis lies in closely analyzing trial completion rates and instances of voluntary withdrawal among these participants.

# Unveiling the Essence of Observational Studies

As a participant in this medical trial, you become an integral part of an observational study, a unique category of clinical trial meticulously crafted to gather insights by observing individuals while keeping their care plans untouched.

Researchers will solely engage in the observation of your journey, meticulously evaluating the outcomes of your condition without any interference. This particular trial design plays a pivotal role in enriching our understanding of the organic evolution of a specific medical condition and its impact on those who bear its diagnosis. By actively engaging in this observational study, you play a dynamic role in propelling the boundaries of medical knowledge and fostering improvements in the care extended to individuals grappling with the same affliction.

# This Trial Compared To Other Metastatic Prostate Cancer Clinical Trials

It is crucial to recognize that the essence of this clinical trial rests upon an observational framework, signifying that your involvement will not encompass the administration of specific treatments or interventions within its scope. However, it is essential to grasp the diverse spectrum of metastatic prostate cancer clinical trials, including interventional trials that entail participants undergoing specific treatment regimens.

Arriving at an informed decision regarding your potential participation in a clinical trial necessitates an active approach of exploration and comparison among diverse studies. A treasure trove of information regarding studies related to metastatic prostate cancer can be accessed through platforms such as clinicaltrials.gov. Moreover, the dedicated online hub by Power presents an exhaustive compilation of ongoing metastatic prostate

<u>cancer clinical trials</u> actively seeking participants. By delving into diligent research and acquiring a holistic understanding of various clinical trial formats, you empower yourself to confidently shape your participation choice.

## Active Participation in Clinical Trial Surveys

In the realm of this observational clinical trial, we extend a heartfelt invitation for you to share your experiences with us. This endeavor entails your periodic completion of questionnaires every two weeks, a commitment that is estimated to require approximately 20-30 minutes of your valuable time. Furthermore, at quarterly intervals, we are prepared to arrange check-in calls, persisting as long as your involvement in the trial continues.

It is of paramount significance to underscore that your engagement in the survey phase of the trial is purely voluntary. The autonomy to decide whether to address specific questions or the entirety of the questionnaire resides entirely with you, and you possess the independence to conclude your participation in the trial whenever you choose. We deeply acknowledge that the decision to partake in a clinical trial is a deeply personal one, and our unwavering commitment is directed towards offering the necessary support. Your privacy and comfort remain steadfast priorities, and we are dedicated to honoring and supporting your decision-making journey throughout the unfolding of the trial.

# Upholding the Secrecy of Your Responses

Maintaining the utmost secrecy of your information remains of paramount importance throughout the entirety of this clinical trial. In order to ensure your anonymity, we kindly advise you to avoid including any personal or identifiable specifics in your questionnaire responses. The devoted research team is steadfast in their commitment to strengthening the safeguard of your confidentiality. Nevertheless, it's important to recognize that specific legal circumstances may arise, necessitating the disclosure of your data.

Potential Hazards

While clinical trials undoubtedly drive medical progress, it is paramount to acknowledge the potential risks to participants' health, particularly in trials exploring novel treatments.

However, our observational clinical trial sets a different course, proactively mitigating these risks by avoiding the introduction of novel interventions to participants. Instead, our primary emphasis revolves around careful observation and outcome measurement, ensuring that unnecessary health hazards are not introduced.

# **Anticipated Benefits**

While immediate benefits may not be readily observable for individuals involved in this observational clinical trial, their engagement has the potential to ripple through the lives of others. The reservoir of data compiled from participants will fuel the refinement of future strategies for enrolling metastatic prostate cancer patients, potentially opening up broader avenues for medical research. By embarking on this clinical expedition, individuals can serve as catalysts for transformative change within the landscape of medical research, potentially reshaping the path for future metastatic prostate cancer patients.

# Navigating the Depths of Clinical Trial Inclusiveness

For those with a keen interest in delving into the intricate landscape of representation in clinical trials, a wealth of online resources eagerly awaits your active participation.

Whether your objective is to unravel challenges and prospects regarding clinical trial diversity, or you simply aim to enrich your personal knowledge, these sources can stand as a guide:

National Academies of Sciences, Engineering, and Medicine. "Improving representation in clinical trials and research: building research equity for women and underrepresented groups." (2022).

Ma, Manuel A., Dora E. Gutiérrez, Joanna M. Frausto, and Wael K. Al-Delaimy. "Minority representation in clinical trials in the United States: trends over the past 25 years." In *Mayo Clinic Proceedings*, vol. 96, no. 1, pp. 264-266. Elsevier, 2021.

### Affirmation of Informed Consent

I affirm that I have dedicated substantial time to comprehensively understand and absorb the contents enclosed within the informed consent form, either through independent review or with the assistance of a trusted individual who has conveyed its essence to me. All inquiries and uncertainties that occupied my thoughts have been thoroughly addressed satisfactorily.

I am acutely aware that my participation in this study is a result of my voluntary decision, and the authority to withdraw my consent rests solely with me, without any obligation to provide a rationale or incur financial obligations. I have been expressly informed that a duplicate of this informed consent form will be provided for my personal documentation.

Having diligently reflected upon and evaluated the entirety of the information presented to me, I hereby provide my concurrence to engage in this study, symbolizing my autonomous choice.

| Printed Name of Participant |
|-----------------------------|
| Participant Signature |
| <br>Date |

Confirmation by Informed Consent Facilitator

I firmly confirm that I have engaged in a comprehensive dialogue with the participant, systematically unraveling the complexities encapsulated within this written document. My objective was to ensure the participant's thorough comprehension of the trial's

overarching objectives, employed methodologies, potential risks and benefits, as well as other essential elements intrinsic to the metastatic prostate cancer clinical trial.

Adequate space was provided to the participant, fostering the emergence of inquiries and facilitating the clarification of uncertainties or misconceptions. It is essential to underscore that the participant's engagement in this trial is a result of their voluntary decision, and they retain the unrestricted prerogative to discontinue their involvement at any point, driven by any rationale, without incurring any financial obligations.

Following the participant's provision of consent, a meticulously preserved duplicate of this written document was provided to them, serving as a repository for their individual records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| Date |